CLINICAL TRIAL: NCT05966571
Title: Ovarian Innervation Study in Patients With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Albanian University (Other)
Responsible Party: Principal Investigator, Elko Gliozheni, Principal Investigator, Albanian University
Other Study IDs: 1576/prot 1
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCOS women: Ovarian biopsy will be performed on PCOS women meeting the inclusion criteria undergoing surgery for other reasons . A sample of the ovarian tissue will be of a few millimeters in size and taken on only one of the ovaries.
  Interventions: Procedure: Ovary Biopsie

INTERVENTIONS:
Procedure: Ovary Biopsie — Ovarian biopsy will be performed on patients meeting the inclusion criteria undergoing surgery for other reasons. Ovarian biopsy will be of a few millimeters in size and taken on only one of the ovaries.

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a complex endocrine disorder characterized by hyperandrogenism, insulin resistance, and ovulatory dysfunction. One of the diagnostic criteria for PCOS is the presence of polycystic ovaries, which are enlarged ovaries with multiple follicles on ultrasound. However, the mechanisms that lead to the development of polycystic ovaries in PCOS are not completely understood. One potential area of investigation is the role of ovarian innervation in the pathophysiology of PCOS. Therefore, the aim of this study is to evaluate the ovarian innervation in PCOS patients through ovarian biopsy sampling.

DETAILED DESCRIPTION:
This is a cross-sectional study that will involve the recruitment of patients diagnosed with PCOS. The study will be conducted at a tertiary care center Koco Gliozheni Maternity, Faculty of Medicine of Tirana, Department of Obstetrics and Gynecology with expertise in gynecology and endocrinology and will then be examined with the aid of the department of Biology and Physiology of the University of Perugia. The study protocol will be approved by the institutional ethics committee, and written informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of PCOS based on the Rotterdam criteria,
* No use of hormonal contraception or medications for at least 3 months prior to the study,
* No history of ovarian cancer.

Exclusion Criteria:

* History of pelvic inflammatory disease or other pelvic infections,
* Use of medications that may affect ovarian function or innervation, such as antipsychotics or antidepressants
* Presence of ovarian cysts > 5 cm on ultrasound

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: PCOS Patients who meet the inclusion criteria will undergo a detailed medical history, physical examination, and laboratory investigations including hormonal evaluation as necessary (testosterone, sex hormone-binding globulin, luteinizing hormone, follicle-stimulating hormone, prolactin, thyroid-stimulating hormone, and cortisol).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Quantify nerve fibers | day 0
  identify and quantify the nerve fibers in the ovarian stroma and follicles
Identifying nerual markers | day 0
  Identification of neural markers such as Protein Gene Product 9.5 (PGP 9.5), by useing antibodies (es. neurotransmitters such as tyrosine hydroxylase (TH), vasoactive intestinal peptide (VIP), and neuropeptide Y).

CONTACTS AND LOCATIONS:
Overall Officials: Elko Gliozheni, Dr, Principal Investigator — University of Medicine
Locations (1):
- University of medicine of Tirana, Tirana, Albania